CLINICAL TRIAL: NCT02387892
Title: Do Vitamin D Fortified Cheese and Yogurt Products Support Vitamin D Status and Functional Outcomes in Young Children? Phase 2
Brief Title: Fortified Cheese and Yogurt Products and Vitamin D Status in Young Children? Phase 2
Acronym: D-KIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HW-14-01-P2
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — Cheese; Yogurt; Vitamin D; Dairy Products; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Cheese & yogurt
  Interventions: Dietary Supplement: Cheese & yogurt
- Treatment (Experimental): Cheese & yogurt + Vitamin D
  Interventions: Dietary Supplement: Cheese & yogurt + Vitamin D

INTERVENTIONS:
Dietary Supplement: Cheese & yogurt + Vitamin D — cheese & yogurt with added 420 IU cholecalciferol
  Other Names: dairy products + cholecalciferol
  Arms: Treatment
Dietary Supplement: Cheese & yogurt — Cheese & yogurt without added vitamin D
  Other Names: dairy products
  Arms: Control

SUMMARY:
This study is being done to test if adding vitamin D to cheese and yogurt products will help children further improve their vitamin D intake. All children will be given a six month supply of the milk products. One group will receive yogurt and cheese products already sold in stores, while the other group will receive yogurt and cheese products with added vitamin D. This will show if milk products with added vitamin D help maintain vitamin D intake and child health.

The investigators are asking children 2 through 8 years old to participate. Children must not have any medical conditions that affect their bones or vitamin D levels. They must not be taking vitamin D supplements or medications that affect bone. This study will last for 6 months. The investigators expect 60 children from the Montreal area will participate in this study.

Children will be randomly placed in one of the two study groups. There will be an equal number of children in each group. All groups will go through the exact same procedures during the study; the only difference between groups will be the amount of vitamin D in the milk products they will consume each day. Families will not know which group their child is in until the study is complete. Children will continue to drink their regular milk at home and the investigators will provide flavoured yogurts and cheese to eat every day for the entire 6 month study. Families will be given a fresh supply of the yogurt or cheese products every 4 weeks along with instructions.

There are 3 study meetings for the parent and child to attend which take place at the Mary Emily Clinical Nutrition Research Unit. The clinic is located on the Macdonald Campus of McGill University in Ste. Anne-de-Bellevue, QC. The first visit is at the start of the study, the second is at the end of 3 months and the last visit is at the end of the 6 month study.

DETAILED DESCRIPTION:
Primary Objective:

1. Establish how much vitamin D intake from food is required to maintain vitamin D status consistent with 75 nmol/L of serum 25(OH)D in all children from the beginning of the UVB-void period (beginning of October) to the end of the winter period (end of April). The amount of vitamin D will be selected based on Phase 1 data (January to April 2014).

   It is hypothesized that total intakes half of the EAR of 400 IU (i.e. 200 IU/d as a typical intake by young children) will result in exceeding a serum 25(OH)D of 40 nmol/L as the population target that aligns with the current EAR value. Intakes reaching the RDA of 600 IU will support serum concentrations of 25(OH)D over 50 nmol/L (and enable further investigations regarding functional outcomes in bone such as BMC and BMD).

   Secondary Objectives:
2. Demonstrate that children with higher vitamin D status (≥ 50 nmol/L 25(OH)D) will have improved biomarkers of bone mineral metabolism compared to those with lower vitamin D status (<50 nmol/L 25(OH)D).

It is hypothesized that children with higher vitamin D status will have lower PTH and CTx with higher P1NP and normal iCa, suggesting that other bone health outcomes would also be improved; in preparation for the follow-up studies.

Design: Parallel randomized controlled study using fortified milk and milk products.

Population: Healthy children (n=60) 2 to 8 y of age from the Greater Montreal Area.

This study uses two groups (based on results from phase 1) to establish how much vitamin D intake from food is required to maintain vitamin D status consistent with 75 nmol/L throughout the duration of winter.

Control Group 1: regular fortified milk + regular cheeses/yogurts Intervention Group 2: regular fortified milk and fortified yogurts and cheeses

Estimated Vitamin D intake from 2.5 servings of Milk and Milk Products and other Foods1 All serving sizes are ½ of a Canada's Food Guide Milk and Alternatives Serving.

Study Group Fluid Milk (2x 125 ml) Yogurt drink (2x93 ml) Cheese (21 g) Other Foods Total/d Dose-response increments

1. (control) 100 IU ~30 IU tr. IU 10-65 IU 140-195 0
2. 100 IU 300 IU 300 IU 10-65 IU 410-465 420 IU vs grp 1

1 Fluid milk servings based on previous data where median intake was 1.7 servings/d [IQR 1.0-2.3]; total of all milk products servings was 2.5 [IQR: 1.7-3.3]; and vitamin D intake from other foods provided ~65 IU/d. All serving sizes are ½ of a Canada's Food Guide Milk and Alternatives Serving. The specially fortified cheeses will be made by Agropur Cooperative, St-Hubert, Quebec and the specially fortified yogurt products will be made by Ultima Foods Inc., Quebec. All products are verified to be within 5% of vitamin D content. The yogurt beverage has 15 IU/93 ml and the fortified product 150 IU/93 ml. The cheese will be standard or made with one fortification level (0 or 300 IU/25 g serving). All serving sizes have been selected based on the target population and typical intakes. There will be no difference in taste between the fortified and non-fortified products.

A 24 h total food intake (day prior to sampling) and validated 1 mo food frequency questionnaire (FFQ) for calcium and vitamin D assessments will be conducted. Nutrient intake will be generated using Nutritionist Pro™ (Axxya Systems LLC, Stafford, TX, US) and the Canadian Nutrient File version 2010b. Compliance is also by monthly telephone survey and unused product.

Demographics, Skin Pigmentation and UVB: Surveys at baseline with parents or legal guardians will be used to estimate socioeconomic status (education and household income). Race will be collected to facilitate understanding of the relationships among culture, skin pigmentation and baseline vitamin D status [5,6]. Data regarding sun exposure during the previous month will be collected as a percentage of body surface area (BSA) exposed frequency of sunscreen use and total hours spent in direct sunlight per day. Sun index will be calculated for each child as necessary (i.e. travel), by multiplying the % BSA exposed by the time spent outside (minutes per day). This index does not consider use of sun block, which is captured by survey in event of travel. Skin type at baseline will be established by measuring pigmentation three times at each site for constitutive pigmentation at the inner upper arm and facultative pigmentation at the forehead, mid-forearm and lower leg using a spectrophotometer (CM-700d/600d, Konica Minolta, Ramsey, NJ, USA).

Anthropometry: Height will be measured using a portable stadiometer (Seca 213, Seca Medical Scales and Measuring Systems, Hamburg, Germany) and body weight measured using a digital scale (Home Collection 63-8711-0, Trileaf Distribution, ON, Canada: calibrated) with the child wearing light clothing and no shoes. Body mass index (BMI) will be calculated. Z-scores for weight, height and BMI will be calculated using the WHO 2007 growth standards/references for children under/over 5 y (WHO AnthroPlus, Geneva, Switzerland). A BMI Z-score of +2 will be considered obese as is important to exclusion criteria; and possibly changes over time.

At baseline and 6 months, dual-energy x-ray absorptiometry (DXA) will be used to quantify total body and regional fat masses. This will be done to help explain any differences in response to vitamin D intakes since more central deposition of adipose tissue relates to vitamin D status in adults [15]. DXA will also be used to measure changes in BMC and BMD over the 6 month period to explore their relationship to vitamin D status. Measurements will be taken using a Hologic 4500A clinical densitometer. Whole body, lumbar spine (L1-4) and forearm scans will be undertaken to measure BMC and BMD, children will wear standardized clothing (pyjama bottoms and T-shirt). The whole body scan technique also provides total body fat, but does not distinguish subcutaneous from visceral fat depots. Abdominal adipose will be estimated using sub-region analysis of the full torso and the between the last rib and the iliac crests. Total body fat (kg and %) and trunk fat (kg) values are available from the DXA software. Although DXA measures of trunk fat mass reflect adipose tissue in subcutaneous and visceral depots, DXA-derived measures agree well with CT in women [16].

To measure volumetric BMD (vBMD) as well as bone architecture, peripheral quantitative computer tomography (pQCT) (XCT-2000; Stratec, Pforzheim, Germany) will be used. pQCT is able to distinguish between type of bone (cortical and trabecular). For the tibia, length of the non-dominant tibia is measured as the distance from the distance between the palpated lateral condyle and the lateral malleolus. Single slices are measured 4% and 66% proximally from the distal end of the tibia. The 4% site will provide a trabecular measurement whilst the 66% site will provide a cortical measurement.

Blood Sampling and Procurement: Fasted (nothing after midnight) venipuncture samples (total 6.5 ml) will be taken ~ 0800 h [17]; breakfast will follow at the research site.

Vitamin D Status and Bone Biomarkers: In serum (from 3 ml whole blood; stored -80°C until analysis), total 25(OH)D (25 µl) as well as PTH will be measured using an immunoassay (Liaison, Diasorin) with proven agreement with LC-MS/MS [20].

ELIGIBILITY:
Inclusion Criteria:

* Children 2 through 8 years of age;
* Healthy body weight for age.

Exclusion Criteria:

* Regular use of vitamin D supplements;
* Lactose intolerant;
* Don't drink milk or eat cheese or yogurt;
* Prior treatment for biochemically confirmed vitamin D deficiency;
* Known or suspected medical conditions associated with bone and vitamin D including rickets, osteomalacia, liver disease, renal disease, immobilization (complete or partial), fractures, and disorders of the parathyroid gland;
* Known or suspected chronic illness of childhood, such as asthma, cancer, Crohn's disease, nephrotic syndrome, rheumatic conditions, and diabetes, etc;
* Use in the past 3 months of medications known to affect bone and/or mineral ion metabolism including oral/systemic/inhaled glucocorticoids, phosphate therapy or vitamin D analogues. Bisphosphonates are also included in this category;
* however, because of their long-half lives and persistence in bone tissue, any prior use of bisphosphonate therapy precludes enrolment;
* Conditions in which the procurement of 8 ml of blood would compromise the health of the patient (i.e. patients with severe anemia).

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Vitamin D serum concentration | 6 month
  How much vitamin D intake from food is required to maintain vitamin D status consistent with 50 nmol/L of serum 25(OH)D in all children from the beginning of the UVB-void period (beginning of October) to the end of the winter period (end of April).

SECONDARY OUTCOMES:
Bone Mineral Density | 6 month
  Demonstrate that children with higher vitamin D status (≥ 50 nmol/L 25(OH)D) will have improved biomarkers of bone mineral metabolism compared to those with lower vitamin D status (<50 nmol/L 25(OH)D).
Bone Mineral Density | 6 month
  Demonstrate that children with higher vitamin D status (≥ 50 nmol/L 25(OH)D) will have improved BMC and BMD compared to those with lower vitamin D status (<50 nmol/L 25(OH)D) using DXA and pQCT.
Body Composition | 6 month
  Examine the effect of higher vitamin D status (≥ 50 nmol/L 25(OH)D) on lean mass compared to those with lower vitamin D status (<50 nmol/L 25(OH)D) using DXA and pQCT.
Body Compositon | 6 month
  Examine the effect of higher vitamin D status (≥ 50 nmol/L 25(OH)D) on fat mass compared to those with lower vitamin D status (<50 nmol/L 25(OH)D) using DXA and pQCT.

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, Principal Investigator — McGill University
Locations (1):
- Mary Emily Clinical Nutrition Research Unit, Sainte-Anne-de-Bellevue, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brett NR, Parks CA, Lavery P, Agellon S, Vanstone CA, Kaufmann M, Jones G, Maguire JL, Rauch F, Weiler HA. Vitamin D status and functional health outcomes in children aged 2-8 y: a 6-mo vitamin D randomized controlled trial. Am J Clin Nutr. 2018 Mar 1;107(3):355-364. doi: 10.1093/ajcn/nqx062. PMID 29566192